CLINICAL TRIAL: NCT03069599
Title: Differential Immunologic Signature After Pancreatic Cancer Treatment: Does Irreversible Electroporation Lead to a Prolonged and Potent T-cell Mediated Immune Response Compared to Surgical Resection?
Brief Title: Immune Response After Pancreatic Cancer Treatment
Acronym: IRE Immuno
Status: Terminated | Type: Observational
Why Stopped: PI left hospital
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-02037
Record Dates: First submitted 2016-12-20; First posted 2017-03-03 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Electroporation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 10 IRE locally advanced: patients undergoing in situ IRE for locally advanced pancreatic
  Interventions: Procedure: irreversible electroporation (IRE)
- 10 IRE borderline resection: patients undergoing margin accentuation IRE for borderline resectable disease
  Interventions: Procedure: irreversible electroporation (IRE)
- 10 resection only: patients undergoing surgical resection only

INTERVENTIONS:
Procedure: irreversible electroporation (IRE) — Irreversible electroporation is an emerging, mainly non-thermal ablative modality. It circumvents some downsides of thermal ablation and has the potential for broad application among patients with pancreatic cancer.
  Groups: 10 IRE borderline resection; 10 IRE locally advanced

SUMMARY:
The aim of this project is to describe the differential immunologic responses of patients who undergo in situ IRE, margin accentuation IRE with surgical resection of the primary tumor, and surgical resection of the primary tumor only. The primary hypothesis is that IRE induces a long and sustained activation of the cell-mediated immune system, which is distinct from the immune response after surgical resection only. The primary endpoint of this study is the comparison of the CD4+/CD8+ ratio as an indicator of antitumor immunity both longitudinally within a group after the intervention and over time between the three groups. CD4+/CD8+ ratio will be measured preoperatively and at postoperative days 1, 7, 42, and 180. As a secondary outcome, additional measurements will be taken to more specifically characterize the immune response based on peripheral blood samples. Flow cytometry will be used to quantify cell subsets, and ELISA will be used to measure cytokine levels , at the same time-points as for the primary outcome. Each group of patients as described above will consist of 10 consecutive pancreatic cancer patients. Patients aged 18 or older with resectable, borderline resectable, or locally advanced pancreatic cancer will be included. Patients with locally advanced disease will undergo 3 months of preoperative chemotherapy with monitoring to exclude metastatic disease. Main exclusion criteria are cardiac conduction abnormalities and signs of distant metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to undergo general anesthesia (ASA ≤ 4)
* Performance status ECOG <=2 (Eastern Cooperative Oncology Group)
* Life expectancy of at least 6 months
* Resectable, borderline resectable, or locally advanced pancreatic cancer
* Patients who have locally advanced disease have to show no tumor progression after 3 month of neo-adjuvant chemotherapy+/-XRT before undergoing in situ IRE

Exclusion Criteria:

* Cardiac AV conduction abnormalities, ventricular fibrillation
* History of epilepsy
* Recent history of myocardial infarction (2 months)
* Evidence of distant metastasis (e.g. liver, lung, peritoneum)
* Informed consent cannot be given by the patient
* Known hypersensitivity to the IRE electrodes (stainless steel 304L)
* Women of childbearing potential who are pregnant, breast feeding, or not taking an adequate method of contraception at the time of procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing an established procedure for pancreatic cancer. The assignment into either group will be independent of this research proposal and rely completely on clinical judgment. Main outcomes will be changes in immunological short-term and long-term outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2020-02-25 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Immunological outcome | 42 days
  flowcytometry
Immunological outcome | 6 months
  Flowcytometry
Immunological outcome | 9 months
  Flowcytometry
Immunological outcome | 42 days
  ELISA
Immunological outcome | 6 months
  ELISA
Immunological outcome | 9 months
  ELISA

SECONDARY OUTCOMES:
Number of local tumor recurrences | 42 days
  measured via CT
Number of local tumor recurrences | 3 months
  measured via CT
Number of local tumor recurrences | 6 months
  measured via CT
Number of local tumor recurrences | 9 months
  measured via CT
Number of distant tumor recurrences | 42 days
  measured via CT
Number of distant tumor recurrences | 3 months
  measured via CT
Number of distant tumor recurrences | 6 months
  measured via CT
Number of distant tumor recurrences | 9 months
  measured via CT
Overall survival | 42 days
  survival of patient
Overall survival | 3 months
  survival of patient
Overall survival | 6 months
  survival of patient
Overall survival | 9 months
  survival of patient
Cancer specific survival | 42 days
  survival of patient
Cancer specific survival | 3 months
  survival of patient
Cancer specific survival | 6 months
  survival of patient
Cancer specific survival | 9 months
  survival of patient

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Worni, MD, Principal Investigator — Inselspital Berne
Locations (1):
- Inselhospital, Bern, Switzerland